CLINICAL TRIAL: NCT05768295
Title: Multicentric Observational Study Confirming the Performance and Safety of the Axiom® BL X3 Implants
Acronym: Prospective_X3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anthogyr (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2101
Record Dates: First submitted 2023-01-27; First posted 2023-03-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Surgical Operation; Edentulous Jaw; Edentulous Mouth; Implant
Keywords: survival rate; success rate; Anthogyr; Axiom® BL X3
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: according to local regulation : The study is an investigation on Medical Device CE marked used in its intended purpose without the objective of CE marking or establishing conformity and with additional procedure non-invasive or non-burdensome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axiom BL X3 (Other): Dental implant Axiom BL X3
  Interventions: Device: Axiom BL X3

INTERVENTIONS:
Device: Axiom BL X3 — collecting data on the use of Axiom BL X3 and patient satisfaction

SUMMARY:
This Post-Market Clinical Follow-Up study aims to document the success and survival of the Axiom® BL X3 Implants up to 3 years after loading.

DETAILED DESCRIPTION:
The total study duration for each patient should be 3 years after loading. .

The investigational devices are CE-(Conformité Européenne, meaning European Conformity) marked product.

14 centers will participate in France

Implants used are Axiom® BL X3 with lengths ranging from 6.5 to 18 mm and diameters ranging from 3.4 to 6.4 mm.

The study and any amendments will be performed as far as possible according to International Organization for Standardization (ISO) 14155, 21CFR 820 for FDA requirement and conform to the Declaration of Helsinki (last revision Fortaleza 2013) and local legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide their informed consent for study participation and must be willing and able to attend control visit (in the standard of care)
* Patients must be males or females who are a minimum of 18 years of age
* Patients seeking an implant supported restoration
* Patient Affiliated to (or beneficiary of) the French Social Security
* Patients who do not present any contraindication for implant restoration, in accordance to IFU

Exclusion Criteria:

* Patients who have no follow-up visit planned with the investigator or co-investigators
* Patients with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance with study visit or unreliability
* A woman who is pregnant or planning to become pregnant at any point during the study duration
* Patients currently participating in another clinical research
* Patients who present contraindication for implant restoration, in accordance to IFU
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Implant success rate | 3 years after loading
  The success rate will be assessed according to the criteria of Buser
  * no detectable clinical mobility (hand testing)
  * no radiolucency surrounding the total surface of the implant
  * no persistent pain refractory to medical therapy
  * no recurrent peri-implant infection

SECONDARY OUTCOMES:
Implant survival rate | 6, 12 months, and 3 years after loading
  A surviving implant is an implant that is in place at the time of evaluation
Prosthesis survival rate | 6, 12 months, and 3 years after loading
  a surviving prosthesis is a prosthesis that is not broken at the time of evaluation
Prosthesis success rate | 6, 12 months, and 3 years after loading
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention during the entire observational period.
Marginal bone level changes | 12 months and 3 years after loading
  Change in crestal bone level measured by analysis of standardized peri-apical xrays [mm]
Patient Reported Outcome | 6, 12 months, and 3 years after loading
  The local language version of the OHIP-14 is a self-reported questionnaire that measures dysfunction, discomfort and disability attributed to oral conditions. The questionnaire focuses on seven dimensions of impact: Functional limitation; Pain; Psychological discomfort; Physical disability; Psychological disability; Social disability; Handicap. The patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4).
Physician satisfaction of the implant stability | at the time of implant placement
  Likert scale : The likert scale will be used for consistency and provides five possible answers to a statement or question that allows respondents to indicate their positive-to-negative strength of agreement or strength of feeling regarding the question or statement.
Interim Implant success rate | 6, 12 months
  A surviving implant is an implant that is in place at the time of evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Margossian, Dr, Principal Investigator — Cabinet Dr Margossian
Locations (13):
- France (13):
  - Cabinet Dentaire Les Aravis, Annecy
  - Cabinet Dr Fumery, Beauvais
  - Cabinet Dr Vigouroux, Cadaujac
  - Cabinet dentaire Octogone, Draguignan
  - Cabinet dentaire Dr Murcia, Le Bouscat
  - Cabinet Dentaire Patrice Margossian, Marseille
  - Cabinet Dr Bruet, Moulins
  - Cabinet Dr Gris, Royan
  - Cabinet Dr Soriano, Saint-Jeoire
  - Cabinet Dr Monnot, Sallanches
  - Cabinet BAG, Toulouse
  - Implantys, Villefranche-sur-Saône
  - Cabinet Dr Broda, Villepreux

IPD SHARING:
Plan to Share IPD: No